CLINICAL TRIAL: NCT06845592
Title: SHARP - Safely Delivered Targeted High-dose Irradiation Followed by Adoptive Immunotherapy with Regulatory and Conventional T Cells to Increase Potency of Hematopoietic Stem Cell Transplantation in High-risk Acute Leukemia
Brief Title: Safely Delivered Targeted High-dose Irradiation Followed by Adoptive Immunotherapy with Regulatory and Conventional T Cells to Increase Potency of Hematopoietic Stem Cell Transplantation in High-risk Acute Leukemia
Acronym: SHARP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Of Perugia (Other)
Responsible Party: Principal Investigator, Antonio Pierini, Principal Investigator, University Of Perugia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHARP
Record Dates: First submitted 2025-02-14; First posted 2025-02-25 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Acute Myeloid Leukaemia (AML); Acute Lymphoblastic Leukemia ALL; High Risk Leukaemia; Leukaemia Relapse
Keywords: AML; ALL; SHARP; Total marrow/lymphoid irradiation; Treg; Tcon; Relapse
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Recurrence | interventions — Lymphatic Irradiation

STUDY DESIGN:
Intervention Model Description: A Simon's Minimax two-stage design has been chosen for predicting number of patients and duration of the study. Such design allows the investigator to early stop patient enrollment in case of unexpected futility.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TMLI based contioning and Treg/Tcon adoptive immunotherapy in allogeneic cell transplantation (Experimental): All enrolled patients will receive a 20Gy-TMLI based conditioning regimen followed by the infusion of donor graft and Treg/Tcon adoptive immunotherapy
  Interventions: Radiation: total marrow/lymphoid irradiation

INTERVENTIONS:
Radiation: total marrow/lymphoid irradiation — Combination of 20 Gy TMLI with Treg/Tcon adoptive immunotherapy in allogeneic cell transplantation

SUMMARY:
The study is a monocentric, interventional study that evaluates the efficacy of allogeneic HLA-matched or haploidentical transplantation consisting of an irradiation-based conditioning regimen coupled with donor Treg/Tcon adoptive immunotherapy for high-risk acute leukemia patients.

ELIGIBILITY:
Inclusion Criteria:

* AML patients

  * Diagnosis of AML with indication to allogeneic hematopoietic cell transplantation.
  * Diagnosis of adverse genetic risk leukemia or presence of MRD or active disease (bone marrow infiltration 5-30%) at the time of the transplant procedure.
  * Availability of a hematopoietic stem cell donor (family or unrelated HLA-matched or HLA-haploidentical with the patient) suitable to be treated with G-CSF (10 mcg/kg/die) for a maximum of 7 days and able to tolerate 2 or more leukaphereses.
  * Age ≥ 18 and ≤ 65 years
  * ECOG ≤ 2
  * HCT-CI ≤ 4 (51,52)
  * Absence of relevant psychiatric diseases
  * Signature of the informed consent

ALL patients

* Diagnosis of ALL, either T or B (Philadelphia negative) or mixed phenotype with indication to allogeneic transplant
* Presence of MRD or active disease (bone marrow infiltration 5-30%) or patient with ≥ 2nd complete hematologic remission at the time of the transplant procedure.
* Availability of a hematopoietic stem cell family donor (family or unrelated HLA-matched or HLA-haploidentical with the patient) suitable to be treated with G-CSF (10 mcg/kg/die) for a maximum of 7 days and able to tolerate 2 or more leukaphereses.
* Age ≥ 18 and ≤ 65 years
* ECOG ≤ 2
* HCT-CI ≤ 4
* Absence of relevant psychiatric diseases
* Signature of the informed consent

Exclusion Criteria:

* AML patients

  * AML in CR MRD-
  * AML with > 5% peripheral blasts or bone marrow infiltration ≥ 30%
  * Age < 18 years or > 65 years
  * ECOG > 2
  * Unacceptable lung, liver, kidney, and/or heart function and presence of relevant psychiatric diseases according to clinical judgment
  * Pregnancy
  * No signature of the informed consent
* ALL patients

  * ALL with > 5% peripheral blasts or bone marrow infiltration ≥30%
  * Philadelphia positive ALL
  * Age < 18 years or > 65 years
  * ECOG > 2
  * Unacceptable lung, liver, kidney, and/or heart function and presence of relevant psychiatric diseases according to clinical judgment
  * Pregnancy
  * No signature of the informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants free from disease 2 years after HSCT | 2 years
  The primary objective of the study is to reduce the incidence of disease relapse after irradiation-based conditioning regimen and Treg/Tcon adoptive immunotherapy-based allogeneic transplantation from HLA-matched or haploidentical donors in high-risk acute leukemia patients.

SECONDARY OUTCOMES:
Number of participants that have reached engraftment 45 days after HSCT | 45 days
  The study will also evaluate the impact of the allogeneic transplantation from HLA-matched or haploidentical donors with irradiation-based conditioning regimen and Treg/Tcon adoptive immunotherapy on major transplantation outcomes in high-risk acute leukemia patients such as full donor type engraftment.
Number of participants that developed grade ≥ 2 acute GvHD | 2 years
  The study will also evaluate the impact of the allogeneic transplantation from HLA-matched or haploidentical donors with irradiation-based conditioning regimen and Treg/Tcon adoptive immunotherapy on major transplantation outcomes in high-risk acute leukemia patients such as grade ≥ 2 acute GvHD.
Number of participants free from chronic GvHD 2 years after HSCT | 2 years
  The study will also evaluate the impact of the allogeneic transplantation from HLA-matched or haploidentical donors with irradiation-based conditioning regimen and Treg/Tcon adoptive immunotherapy on major transplantation outcomes in high-risk acute leukemia patients such as chronic GvHD.

CONTACTS AND LOCATIONS:
Locations (1):
- Università degli Studi di Perugia, Perugia, PG, Italy

REFERENCES:
- [Background] Cordonnier C, Einarsdottir S, Cesaro S, Di Blasi R, Mikulska M, Rieger C, de Lavallade H, Gallo G, Lehrnbecher T, Engelhard D, Ljungman P; European Conference on Infections in Leukaemia group. Vaccination of haemopoietic stem cell transplant recipients: guidelines of the 2017 European Conference on Infections in Leukaemia (ECIL 7). Lancet Infect Dis. 2019 Jun;19(6):e200-e212. doi: 10.1016/S1473-3099(18)30600-5. Epub 2019 Feb 8. PMID 30744963
- [Background] El Fakih R, Hashmi SK, Ciurea SO, Luznik L, Gale RP, Aljurf M. Post-transplant cyclophosphamide use in matched HLA donors: a review of literature and future application. Bone Marrow Transplant. 2020 Jan;55(1):40-47. doi: 10.1038/s41409-019-0547-8. Epub 2019 May 14. PMID 31089284
- [Background] Patil S, Potter V, Mohty M. Review of conditioning regimens for haplo-identical donor transplants using post-transplant cyclophosphamide in recipients of G-CSF mobilised peripheral stem cell. Cancer Treat Rev. 2020 Sep;89:102071. doi: 10.1016/j.ctrv.2020.102071. Epub 2020 Jul 15. PMID 32717620
- [Background] Chistolini P, Cossu G, De Luca M, Marazzi M, Mavilio F, Migliaccio G, et al. LINEE GUIDA PER L'INGEGNERIA DEI TESSUTI E LA TERAPIA CELLULARE. Not DellIstituto Super Sanità. 1999 May 1;Vol. 12:1-8
- [Background] Stern M, Ruggeri L, Mancusi A, Bernardo ME, de Angelis C, Bucher C, Locatelli F, Aversa F, Velardi A. Survival after T cell-depleted haploidentical stem cell transplantation is improved using the mother as donor. Blood. 2008 Oct 1;112(7):2990-5. doi: 10.1182/blood-2008-01-135285. Epub 2008 May 20. PMID 18492955
- [Background] Ruggeri L, Capanni M, Urbani E, Perruccio K, Shlomchik WD, Tosti A, Posati S, Rogaia D, Frassoni F, Aversa F, Martelli MF, Velardi A. Effectiveness of donor natural killer cell alloreactivity in mismatched hematopoietic transplants. Science. 2002 Mar 15;295(5562):2097-100. doi: 10.1126/science.1068440. PMID 11896281
- [Background] Ciurea SO, Cao K, Fernandez-Vina M, Kongtim P, Malki MA, Fuchs E, Luznik L, Huang XJ, Ciceri F, Locatelli F, Aversa F, Castagna L, Bacigalupo A, Martelli M, Blaise D, Handgretinger R, Roy DC, O'Donnell P, Bashey A, Lazarus HM, Ballen K, Savani BN, Mohty M, Nagler A. The European Society for Blood and Marrow Transplantation (EBMT) Consensus Guidelines for the Detection and Treatment of Donor-specific Anti-HLA Antibodies (DSA) in Haploidentical Hematopoietic Cell Transplantation. Bone Marrow Transplant. 2018 May;53(5):521-534. doi: 10.1038/s41409-017-0062-8. Epub 2018 Jan 15. PMID 29335625
- [Background] van der Velden VH, Panzer-Grumayer ER, Cazzaniga G, Flohr T, Sutton R, Schrauder A, Basso G, Schrappe M, Wijkhuijs JM, Konrad M, Bartram CR, Masera G, Biondi A, van Dongen JJ. Optimization of PCR-based minimal residual disease diagnostics for childhood acute lymphoblastic leukemia in a multi-center setting. Leukemia. 2007 Apr;21(4):706-13. doi: 10.1038/sj.leu.2404535. Epub 2007 Feb 8. PMID 17287857
- [Background] van der Velden VH, Cazzaniga G, Schrauder A, Hancock J, Bader P, Panzer-Grumayer ER, Flohr T, Sutton R, Cave H, Madsen HO, Cayuela JM, Trka J, Eckert C, Foroni L, Zur Stadt U, Beldjord K, Raff T, van der Schoot CE, van Dongen JJ; European Study Group on MRD detection in ALL (ESG-MRD-ALL). Analysis of minimal residual disease by Ig/TCR gene rearrangements: guidelines for interpretation of real-time quantitative PCR data. Leukemia. 2007 Apr;21(4):604-11. doi: 10.1038/sj.leu.2404586. Epub 2007 Feb 8. PMID 17287850
- [Background] Elia L, Mancini M, Moleti L, Meloni G, Buffolino S, Krampera M, De Rossi G, Foa R, Cimino G. A multiplex reverse transcriptase-polymerase chain reaction strategy for the diagnostic molecular screening of chimeric genes: a clinical evaluation on 170 patients with acute lymphoblastic leukemia. Haematologica. 2003 Mar;88(3):275-9. PMID 12651265
- [Background] Pierce E, Mautner B, Mort J, Blewett A, Morris A, Keng M, El Chaer F. MRD in ALL: Optimization and Innovations. Curr Hematol Malig Rep. 2022 Aug;17(4):69-81. doi: 10.1007/s11899-022-00664-6. Epub 2022 May 26. PMID 35616771
- [Background] Jung SH, Lee T, Kim K, George SL. Admissible two-stage designs for phase II cancer clinical trials. Stat Med. 2004 Feb 28;23(4):561-9. doi: 10.1002/sim.1600. PMID 14755389
- [Background] Simon R. Optimal two-stage designs for phase II clinical trials. Control Clin Trials. 1989 Mar;10(1):1-10. doi: 10.1016/0197-2456(89)90015-9. PMID 2702835
- [Background] Sorror ML, Maris MB, Storb R, Baron F, Sandmaier BM, Maloney DG, Storer B. Hematopoietic cell transplantation (HCT)-specific comorbidity index: a new tool for risk assessment before allogeneic HCT. Blood. 2005 Oct 15;106(8):2912-9. doi: 10.1182/blood-2005-05-2004. Epub 2005 Jun 30. PMID 15994282
- [Background] Duarte RF, Labopin M, Bader P, Basak GW, Bonini C, Chabannon C, Corbacioglu S, Dreger P, Dufour C, Gennery AR, Kuball J, Lankester AC, Lanza F, Montoto S, Nagler A, Peffault de Latour R, Snowden JA, Styczynski J, Yakoub-Agha I, Kroger N, Mohty M; European Society for Blood and Marrow Transplantation (EBMT). Indications for haematopoietic stem cell transplantation for haematological diseases, solid tumours and immune disorders: current practice in Europe, 2019. Bone Marrow Transplant. 2019 Oct;54(10):1525-1552. doi: 10.1038/s41409-019-0516-2. Epub 2019 Apr 5. PMID 30953028
- [Background] Jagasia MH, Greinix HT, Arora M, Williams KM, Wolff D, Cowen EW, Palmer J, Weisdorf D, Treister NS, Cheng GS, Kerr H, Stratton P, Duarte RF, McDonald GB, Inamoto Y, Vigorito A, Arai S, Datiles MB, Jacobsohn D, Heller T, Kitko CL, Mitchell SA, Martin PJ, Shulman H, Wu RS, Cutler CS, Vogelsang GB, Lee SJ, Pavletic SZ, Flowers ME. National Institutes of Health Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-versus-Host Disease: I. The 2014 Diagnosis and Staging Working Group report. Biol Blood Marrow Transplant. 2015 Mar;21(3):389-401.e1. doi: 10.1016/j.bbmt.2014.12.001. Epub 2014 Dec 18. PMID 25529383
- [Background] Cahn JY, Klein JP, Lee SJ, Milpied N, Blaise D, Antin JH, Leblond V, Ifrah N, Jouet JP, Loberiza F, Ringden O, Barrett AJ, Horowitz MM, Socie G; Societe Francaise de Greffe de Moelle et Therapie Cellulaire; Dana Farber Cancer Institute; International Bone Marrow Transplant Registry. Prospective evaluation of 2 acute graft-versus-host (GVHD) grading systems: a joint Societe Francaise de Greffe de Moelle et Therapie Cellulaire (SFGM-TC), Dana Farber Cancer Institute (DFCI), and International Bone Marrow Transplant Registry (IBMTR) prospective study. Blood. 2005 Aug 15;106(4):1495-500. doi: 10.1182/blood-2004-11-4557. Epub 2005 May 5. PMID 15878974
- [Background] Glucksberg H, Storb R, Fefer A, Buckner CD, Neiman PE, Clift RA, Lerner KG, Thomas ED. Clinical manifestations of graft-versus-host disease in human recipients of marrow from HL-A-matched sibling donors. Transplantation. 1974 Oct;18(4):295-304. doi: 10.1097/00007890-197410000-00001. No abstract available. PMID 4153799
- [Background] Jabbour E, Haddad FG, Short NJ, Kantarjian H. Treatment of Adults With Philadelphia Chromosome-Positive Acute Lymphoblastic Leukemia-From Intensive Chemotherapy Combinations to Chemotherapy-Free Regimens: A Review. JAMA Oncol. 2022 Sep 1;8(9):1340-1348. doi: 10.1001/jamaoncol.2022.2398. PMID 35834222
- [Background] Foa R, Bassan R, Vitale A, Elia L, Piciocchi A, Puzzolo MC, Canichella M, Viero P, Ferrara F, Lunghi M, Fabbiano F, Bonifacio M, Fracchiolla N, Di Bartolomeo P, Mancino A, De Propris MS, Vignetti M, Guarini A, Rambaldi A, Chiaretti S; GIMEMA Investigators. Dasatinib-Blinatumomab for Ph-Positive Acute Lymphoblastic Leukemia in Adults. N Engl J Med. 2020 Oct 22;383(17):1613-1623. doi: 10.1056/NEJMoa2016272. PMID 33085860
- [Background] Couturier MA, Thomas X, Raffoux E, Huguet F, Berthon C, Simand C, Gallego-Hernanz MP, Hicheri Y, Hunault Berger M, Saillard C, Leguay T, Loiseau C, Bene MC, Chevallier P. Blinatumomab + ponatinib for relapsed/refractory Philadelphia chromosome-positive acute lymphoblastic leukemia in adults. Leuk Lymphoma. 2021 Mar;62(3):620-629. doi: 10.1080/10428194.2020.1844198. Epub 2020 Nov 6. PMID 33153370
- [Background] Greil C, Engelhardt M, Ihorst G, Duque-Afonso J, Shoumariyeh K, Bertz H, Marks R, Zeiser R, Duyster J, Finke J, Wasch R. Prognostic factors for survival after allogeneic transplantation in acute lymphoblastic leukemia. Bone Marrow Transplant. 2021 Apr;56(4):841-852. doi: 10.1038/s41409-020-01101-z. Epub 2020 Oct 31. PMID 33130821
- [Background] Srour SA, Milton DR, Bashey A, Karduss-Urueta A, Al Malki MM, Romee R, Solomon S, Nademanee A, Brown S, Slade M, Perez R, Rondon G, Forman SJ, Champlin RE, Kebriaei P, Ciurea SO. Haploidentical Transplantation with Post-Transplantation Cyclophosphamide for High-Risk Acute Lymphoblastic Leukemia. Biol Blood Marrow Transplant. 2017 Feb;23(2):318-324. doi: 10.1016/j.bbmt.2016.11.008. Epub 2016 Nov 14. PMID 27856368
- [Background] Kaito S, Kurosawa S, Najima Y, Sakaida E, Shingai N, Fukuda T, Tachibana T, Uchida N, Ozawa Y, Sawa M, Nakazawa H, Ota S, Kato J, Nakamae H, Katayama Y, Eto T, Tanaka J, Kanda Y, Atsuta Y, Arai Y, Kako S; Adult Acute Lymphoblastic Leukemia Working Group of the Japan Society for Hematopoietic Cell Transplantation. Allogeneic Hematopoietic Stem Cell Transplantation for Adult Philadelphia Chromosome-Negative B-Cell Acute Lymphoblastic Leukemia in Second Complete Remission. Transplant Cell Ther. 2022 Jun;28(6):326.e1-326.e10. doi: 10.1016/j.jtct.2022.03.017. Epub 2022 Mar 17. PMID 35306218
- [Background] Ladbury C, Somlo G, Dagis A, Yang D, Armenian S, Song JY, Sahebi F, Spielberger R, Popplewell L, Parker P, Forman S, Snyder D, Rincon A, Liu A, Frankel P, Wong J. Long-Term Follow-Up of Multiple Myeloma Patients Treated with Tandem Autologous Transplantation Following Melphalan and Upon Recovery, Total Marrow Irradiation. Transplant Cell Ther. 2022 Jul;28(7):367.e1-367.e9. doi: 10.1016/j.jtct.2022.04.022. Epub 2022 May 6. PMID 35534000
- [Background] Jensen LG, Stiller T, Wong JYC, Palmer J, Stein A, Rosenthal J. Total Marrow Lymphoid Irradiation/Fludarabine/ Melphalan Conditioning for Allogeneic Hematopoietic Cell Transplantation. Biol Blood Marrow Transplant. 2018 Feb;24(2):301-307. doi: 10.1016/j.bbmt.2017.09.019. Epub 2017 Oct 12. PMID 29032268
- [Background] Al Malki MM, Palmer J, Tsai NC, Mokhtari S, Hui S, Tsai W, Aldoss I, Ali H, Aribi A, Cao T, Mei M, Sandhu KS, Siddiqi T, Forman SJ, Nakamura R, Marcucci G, Stein A, Wong JYC, Rosenthal J. Total marrow and lymphoid irradiation as conditioning in haploidentical transplant with posttransplant cyclophosphamide. Blood Adv. 2022 Jul 26;6(14):4098-4106. doi: 10.1182/bloodadvances.2022007264. PMID 35838754
- [Background] Stein AS, Al Malki MM, Yang D, Palmer JM, Tsai NC, Aldoss I, Ali H, Aribi A, Artz A, Dandapani S, Farol L, Hui S, Liu A, Nakamura R, Pullarkat V, Radany E, Rosenthal J, Salhotra A, Sanchez JF, Spielberger R, Marcucci G, Forman SJ, Wong J. Total Marrow and Lymphoid Irradiation with Post-Transplantation Cyclophosphamide for Patients with AML in Remission. Transplant Cell Ther. 2022 Jul;28(7):368.e1-368.e7. doi: 10.1016/j.jtct.2022.03.025. Epub 2022 Apr 6. PMID 35398328
- [Background] Stein A, Palmer J, Tsai NC, Al Malki MM, Aldoss I, Ali H, Aribi A, Farol L, Karanes C, Khaled S, Liu A, O'Donnell M, Parker P, Pawlowska A, Pullarkat V, Radany E, Rosenthal J, Sahebi F, Salhotra A, Sanchez JF, Schultheiss T, Spielberger R, Thomas SH, Snyder D, Nakamura R, Marcucci G, Forman SJ, Wong J. Phase I Trial of Total Marrow and Lymphoid Irradiation Transplantation Conditioning in Patients with Relapsed/Refractory Acute Leukemia. Biol Blood Marrow Transplant. 2017 Apr;23(4):618-624. doi: 10.1016/j.bbmt.2017.01.067. Epub 2017 Jan 10. PMID 28087456
- [Background] Heuser M, Freeman SD, Ossenkoppele GJ, Buccisano F, Hourigan CS, Ngai LL, Tettero JM, Bachas C, Baer C, Bene MC, Bucklein V, Czyz A, Denys B, Dillon R, Feuring-Buske M, Guzman ML, Haferlach T, Han L, Herzig JK, Jorgensen JL, Kern W, Konopleva MY, Lacombe F, Libura M, Majchrzak A, Maurillo L, Ofran Y, Philippe J, Plesa A, Preudhomme C, Ravandi F, Roumier C, Subklewe M, Thol F, van de Loosdrecht AA, van der Reijden BA, Venditti A, Wierzbowska A, Valk PJM, Wood BL, Walter RB, Thiede C, Dohner K, Roboz GJ, Cloos J. 2021 Update on MRD in acute myeloid leukemia: a consensus document from the European LeukemiaNet MRD Working Party. Blood. 2021 Dec 30;138(26):2753-2767. doi: 10.1182/blood.2021013626. PMID 34724563
- [Background] DeFilipp Z, Advani AS, Bachanova V, Cassaday RD, Deangelo DJ, Kebriaei P, Rowe JM, Seftel MD, Stock W, Tallman MS, Fanning S, Inamoto Y, Kansagra A, Johnston L, Nagler A, Sauter CS, Savani BN, Perales MA, Carpenter PA, Larson RA, Weisdorf D. Hematopoietic Cell Transplantation in the Treatment of Adult Acute Lymphoblastic Leukemia: Updated 2019 Evidence-Based Review from the American Society for Transplantation and Cellular Therapy. Biol Blood Marrow Transplant. 2019 Nov;25(11):2113-2123. doi: 10.1016/j.bbmt.2019.08.014. Epub 2019 Aug 22. PMID 31446198
- [Background] Giebel S, Marks DI, Boissel N, Baron F, Chiaretti S, Ciceri F, Cornelissen JJ, Doubek M, Esteve J, Fielding A, Foa R, Gorin NC, Gokbuget N, Hallbook H, Hoelzer D, Paravichnikova E, Ribera JM, Savani B, Rijneveld AW, Schmid C, Wartiovaara-Kautto U, Mohty M, Nagler A, Dombret H. Hematopoietic stem cell transplantation for adults with Philadelphia chromosome-negative acute lymphoblastic leukemia in first remission: a position statement of the European Working Group for Adult Acute Lymphoblastic Leukemia (EWALL) and the Acute Leukemia Working Party of the European Society for Blood and Marrow Transplantation (EBMT). Bone Marrow Transplant. 2019 Jun;54(6):798-809. doi: 10.1038/s41409-018-0373-4. Epub 2018 Nov 1. PMID 30385870
- [Background] Dohner H, Wei AH, Appelbaum FR, Craddock C, DiNardo CD, Dombret H, Ebert BL, Fenaux P, Godley LA, Hasserjian RP, Larson RA, Levine RL, Miyazaki Y, Niederwieser D, Ossenkoppele G, Rollig C, Sierra J, Stein EM, Tallman MS, Tien HF, Wang J, Wierzbowska A, Lowenberg B. Diagnosis and management of AML in adults: 2022 recommendations from an international expert panel on behalf of the ELN. Blood. 2022 Sep 22;140(12):1345-1377. doi: 10.1182/blood.2022016867. PMID 35797463
- [Background] Blume KG, Kopecky KJ, Henslee-Downey JP, Forman SJ, Stiff PJ, LeMaistre CF, Appelbaum FR. A prospective randomized comparison of total body irradiation-etoposide versus busulfan-cyclophosphamide as preparatory regimens for bone marrow transplantation in patients with leukemia who were not in first remission: a Southwest Oncology Group study. Blood. 1993 Apr 15;81(8):2187-93. PMID 8471778
- [Background] Forman SJ, Rowe JM. The myth of the second remission of acute leukemia in the adult. Blood. 2013 Feb 14;121(7):1077-82. doi: 10.1182/blood-2012-08-234492. Epub 2012 Dec 14. PMID 23243288
- [Background] Aldoss I, Yang D, Malki MMA, Mei M, Mokhtari S, Artz A, Cao T, Salhotra A, Ali H, Aribi A, Khaled S, Arslan S, Sandhu K, Koller P, Mansour J, Spielberger R, Stein A, Snyder D, Marcucci G, Forman SJ, Nakamura R, Pullarkat V. Allogeneic Hematopoietic Cell Transplantation for Relapsed and Refractory Philadelphia Negative B Cell ALL in the Era of Novel Salvage Therapies. Transplant Cell Ther. 2021 Mar;27(3):255.e1-255.e9. doi: 10.1016/j.jtct.2020.12.020. Epub 2020 Dec 22. PMID 33781525
- [Background] Logan AC. Measurable residual disease in acute lymphoblastic leukemia: How low is low enough? Best Pract Res Clin Haematol. 2022 Dec;35(4):101407. doi: 10.1016/j.beha.2022.101407. Epub 2022 Oct 29. PMID 36517126
- [Background] Thol F, Gabdoulline R, Liebich A, Klement P, Schiller J, Kandziora C, Hambach L, Stadler M, Koenecke C, Flintrop M, Pankratz M, Wichmann M, Neziri B, Buttner K, Heida B, Klesse S, Chaturvedi A, Kloos A, Gohring G, Schlegelberger B, Gaidzik VI, Bullinger L, Fiedler W, Heim A, Hamwi I, Eder M, Krauter J, Schlenk RF, Paschka P, Dohner K, Dohner H, Ganser A, Heuser M. Measurable residual disease monitoring by NGS before allogeneic hematopoietic cell transplantation in AML. Blood. 2018 Oct 18;132(16):1703-1713. doi: 10.1182/blood-2018-02-829911. Epub 2018 Sep 6. PMID 30190321
- [Background] Selove W, Hutchinson L, Makarenko V, Meng X, Tomaszewicz K, Ramanathan M, Cerny J, Nath R, Chen B, Woda B, Bledsoe JR. Impact of pretransplant mutation status on survival after allogeneic stem cell transplant for acute myeloid leukemia. EJHaem. 2021 Jul 22;2(3):514-519. doi: 10.1002/jha2.260. eCollection 2021 Aug. No abstract available. PMID 35844698
- [Background] Buckley SA, Wood BL, Othus M, Hourigan CS, Ustun C, Linden MA, DeFor TE, Malagola M, Anthias C, Valkova V, Kanakry CG, Gruhn B, Buccisano F, Devine B, Walter RB. Minimal residual disease prior to allogeneic hematopoietic cell transplantation in acute myeloid leukemia: a meta-analysis. Haematologica. 2017 May;102(5):865-873. doi: 10.3324/haematol.2016.159343. Epub 2017 Jan 25. PMID 28126965
- [Background] Czyz A, Nagler A. The Role of Measurable Residual Disease (MRD) in Hematopoietic Stem Cell Transplantation for Hematological Malignancies Focusing on Acute Leukemia. Int J Mol Sci. 2019 Oct 28;20(21):5362. doi: 10.3390/ijms20215362. PMID 31661875
- [Background] Lussana F, Caprioli C, Stefanoni P, Pavoni C, Spinelli O, Buklijas K, Michelato A, Borleri G, Algarotti A, Mico C, Grassi A, Intermesoli T, Rambaldi A. Molecular Detection of Minimal Residual Disease before Allogeneic Stem Cell Transplantation Predicts a High Incidence of Early Relapse in Adult Patients with NPM1 Positive Acute Myeloid Leukemia. Cancers (Basel). 2019 Sep 28;11(10):1455. doi: 10.3390/cancers11101455. PMID 31569375
- [Background] Press RD, Eickelberg G, Froman A, Yang F, Stentz A, Flatley EM, Fan G, Lim JY, Meyers G, Maziarz RT, Cook RJ. Next-generation sequencing-defined minimal residual disease before stem cell transplantation predicts acute myeloid leukemia relapse. Am J Hematol. 2019 Aug;94(8):902-912. doi: 10.1002/ajh.25514. Epub 2019 Jun 14. PMID 31124175
- [Background] Araki D, Wood BL, Othus M, Radich JP, Halpern AB, Zhou Y, Mielcarek M, Estey EH, Appelbaum FR, Walter RB. Allogeneic Hematopoietic Cell Transplantation for Acute Myeloid Leukemia: Time to Move Toward a Minimal Residual Disease-Based Definition of Complete Remission? J Clin Oncol. 2016 Feb 1;34(4):329-36. doi: 10.1200/JCO.2015.63.3826. Epub 2015 Dec 14. PMID 26668349
- [Background] Pierini A, Ruggeri L, Saldi S, Tricarico S, Marzuttini F, Viglione V, et al. HLA-Matched Treg/Tcon Allogeneic Hematopoietic Cell Transplantation Is Safe and Ensures Remarkable Chronic GvHD/Leukemia Free Survival in High-Risk Leukemia Patients. Blood. 2022 Nov 15;140(Supplement 1):2133-4
- [Background] Rosenthal J, Wong J, Stein A, Qian D, Hitt D, Naeem H, Dagis A, Thomas SH, Forman S. Phase 1/2 trial of total marrow and lymph node irradiation to augment reduced-intensity transplantation for advanced hematologic malignancies. Blood. 2011 Jan 6;117(1):309-15. doi: 10.1182/blood-2010-06-288357. Epub 2010 Sep 28. PMID 20876852
- [Background] Ferrara JL, Levine JE, Reddy P, Holler E. Graft-versus-host disease. Lancet. 2009 May 2;373(9674):1550-61. doi: 10.1016/S0140-6736(09)60237-3. Epub 2009 Mar 11. PMID 19282026
- [Background] Koreth J, Matsuoka K, Kim HT, McDonough SM, Bindra B, Alyea EP 3rd, Armand P, Cutler C, Ho VT, Treister NS, Bienfang DC, Prasad S, Tzachanis D, Joyce RM, Avigan DE, Antin JH, Ritz J, Soiffer RJ. Interleukin-2 and regulatory T cells in graft-versus-host disease. N Engl J Med. 2011 Dec 1;365(22):2055-66. doi: 10.1056/NEJMoa1108188. PMID 22129252
- [Background] Kennedy-Nasser AA, Ku S, Castillo-Caro P, Hazrat Y, Wu MF, Liu H, Melenhorst J, Barrett AJ, Ito S, Foster A, Savoldo B, Yvon E, Carrum G, Ramos CA, Krance RA, Leung K, Heslop HE, Brenner MK, Bollard CM. Ultra low-dose IL-2 for GVHD prophylaxis after allogeneic hematopoietic stem cell transplantation mediates expansion of regulatory T cells without diminishing antiviral and antileukemic activity. Clin Cancer Res. 2014 Apr 15;20(8):2215-25. doi: 10.1158/1078-0432.CCR-13-3205. Epub 2014 Feb 26. PMID 24573552
- [Background] Hadjis AD, Nunes NS, Khan SM, Fletcher RE, Pohl AP, Venzon DJ, Eckhaus MA, Kanakry CG. Post-Transplantation Cyclophosphamide Uniquely Restrains Alloreactive CD4+ T-Cell Proliferation and Differentiation After Murine MHC-Haploidentical Hematopoietic Cell Transplantation. Front Immunol. 2022 Feb 15;13:796349. doi: 10.3389/fimmu.2022.796349. eCollection 2022. PMID 35242129
- [Background] Nunes NS, Kanakry CG. Mechanisms of Graft-versus-Host Disease Prevention by Post-transplantation Cyclophosphamide: An Evolving Understanding. Front Immunol. 2019 Nov 29;10:2668. doi: 10.3389/fimmu.2019.02668. eCollection 2019. PMID 31849930
- [Background] Ganguly S, Ross DB, Panoskaltsis-Mortari A, Kanakry CG, Blazar BR, Levy RB, Luznik L. Donor CD4+ Foxp3+ regulatory T cells are necessary for posttransplantation cyclophosphamide-mediated protection against GVHD in mice. Blood. 2014 Sep 25;124(13):2131-41. doi: 10.1182/blood-2013-10-525873. Epub 2014 Aug 18. PMID 25139358
- [Background] Kanakry CG, Ganguly S, Zahurak M, Bolanos-Meade J, Thoburn C, Perkins B, Fuchs EJ, Jones RJ, Hess AD, Luznik L. Aldehyde dehydrogenase expression drives human regulatory T cell resistance to posttransplantation cyclophosphamide. Sci Transl Med. 2013 Nov 13;5(211):211ra157. doi: 10.1126/scitranslmed.3006960. PMID 24225944
- [Background] Pierini A, Ruggeri L, Carotti A, Falzetti F, Saldi S, Terenzi A, Zucchetti C, Ingrosso G, Zei T, Iacucci Ostini R, Piccinelli S, Bonato S, Tricarico S, Mancusi A, Ciardelli S, Limongello R, Merluzzi M, Di Ianni M, Tognellini R, Minelli O, Mecucci C, Martelli MP, Falini B, Martelli MF, Aristei C, Velardi A. Haploidentical age-adapted myeloablative transplant and regulatory and effector T cells for acute myeloid leukemia. Blood Adv. 2021 Mar 9;5(5):1199-1208. doi: 10.1182/bloodadvances.2020003739. PMID 33646302
- [Background] Martelli MF, Di Ianni M, Ruggeri L, Falzetti F, Carotti A, Terenzi A, Pierini A, Massei MS, Amico L, Urbani E, Del Papa B, Zei T, Iacucci Ostini R, Cecchini D, Tognellini R, Reisner Y, Aversa F, Falini B, Velardi A. HLA-haploidentical transplantation with regulatory and conventional T-cell adoptive immunotherapy prevents acute leukemia relapse. Blood. 2014 Jul 24;124(4):638-44. doi: 10.1182/blood-2014-03-564401. Epub 2014 Jun 12. PMID 24923299
- [Background] Di Ianni M, Falzetti F, Carotti A, Terenzi A, Castellino F, Bonifacio E, Del Papa B, Zei T, Ostini RI, Cecchini D, Aloisi T, Perruccio K, Ruggeri L, Balucani C, Pierini A, Sportoletti P, Aristei C, Falini B, Reisner Y, Velardi A, Aversa F, Martelli MF. Tregs prevent GVHD and promote immune reconstitution in HLA-haploidentical transplantation. Blood. 2011 Apr 7;117(14):3921-8. doi: 10.1182/blood-2010-10-311894. Epub 2011 Feb 3. PMID 21292771
- [Background] Pierini A, Colonna L, Alvarez M, Schneidawind D, Nishikii H, Baker J, Pan Y, Florek M, Kim BS, Negrin RS. Donor Requirements for Regulatory T Cell Suppression of Murine Graft-versus-Host Disease. J Immunol. 2015 Jul 1;195(1):347-55. doi: 10.4049/jimmunol.1402861. Epub 2015 May 20. PMID 25994967
- [Background] Nguyen VH, Zeiser R, Dasilva DL, Chang DS, Beilhack A, Contag CH, Negrin RS. In vivo dynamics of regulatory T-cell trafficking and survival predict effective strategies to control graft-versus-host disease following allogeneic transplantation. Blood. 2007 Mar 15;109(6):2649-56. doi: 10.1182/blood-2006-08-044529. Epub 2006 Nov 9. PMID 17095616
- [Background] Edinger M, Hoffmann P, Ermann J, Drago K, Fathman CG, Strober S, Negrin RS. CD4+CD25+ regulatory T cells preserve graft-versus-tumor activity while inhibiting graft-versus-host disease after bone marrow transplantation. Nat Med. 2003 Sep;9(9):1144-50. doi: 10.1038/nm915. Epub 2003 Aug 17. PMID 12925844
- [Background] Wing JB, Tanaka A, Sakaguchi S. Human FOXP3+ Regulatory T Cell Heterogeneity and Function in Autoimmunity and Cancer. Immunity. 2019 Feb 19;50(2):302-316. doi: 10.1016/j.immuni.2019.01.020. PMID 30784578
- [Background] Mancusi A, Ruggeri L, Velardi A. Haploidentical hematopoietic transplantation for the cure of leukemia: from its biology to clinical translation. Blood. 2016 Dec 8;128(23):2616-2623. doi: 10.1182/blood-2016-07-730564. Epub 2016 Oct 3. PMID 27697774
- [Background] Aversa F, Tabilio A, Terenzi A, Velardi A, Falzetti F, Giannoni C, Iacucci R, Zei T, Martelli MP, Gambelunghe C, et al. Successful engraftment of T-cell-depleted haploidentical "three-loci" incompatible transplants in leukemia patients by addition of recombinant human granulocyte colony-stimulating factor-mobilized peripheral blood progenitor cells to bone marrow inoculum. Blood. 1994 Dec 1;84(11):3948-55. PMID 7524753
- [Background] Aversa F, Tabilio A, Velardi A, Cunningham I, Terenzi A, Falzetti F, Ruggeri L, Barbabietola G, Aristei C, Latini P, Reisner Y, Martelli MF. Treatment of high-risk acute leukemia with T-cell-depleted stem cells from related donors with one fully mismatched HLA haplotype. N Engl J Med. 1998 Oct 22;339(17):1186-93. doi: 10.1056/NEJM199810223391702. PMID 9780338